CLINICAL TRIAL: NCT06420726
Title: The Feasibility and Acceptability of Resistance Training and Creatine Supplementation to Promote Physical Function in Sarcopenic Colorectal Cancer Survivors
Brief Title: Resistance Exercise and Creatine in Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Ciaran Fairman, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00127362
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Two-arm Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + Creatine (Experimental): 3 days a week of resistance exercise for 10-weeks + 5g day of creatine monohydrate supplementation
  Interventions: Behavioral: Resistance Exercise
- Exercise + Placebo (Placebo Comparator): 3 days a week of resistance exercise for 10-weeks + 5g day of placebo (dextrose supplementation
  Interventions: Behavioral: Resistance Exercise

INTERVENTIONS:
Behavioral: Resistance Exercise — Supervised resistance exercise

SUMMARY:
skeletal muscle mass and function, is prevalent in up to 60% of colorectal cancer patients. This condition arises from a combination of factors such as aging, inactivity, treatment side effects, malnutrition, tumor burden, and inflammation. Given this complexity, singular interventions may not be sufficient to address sarcopenia in this group.

Creatine monohydrate, a compound vital for energy during exercise, has been extensively researched and proven safe and effective across various demographics, including older adults and clinical populations. Studies show that creatine enhances benefits from resistance training, indicating potential to counter muscle mass and function decline post-cancer treatment.

This study aims to assess the feasibilty of combining creatine supplementation with resistance training versus resistance training alone in sarcopenic colorectal cancer survivors. A randomized controlled pilot trial will compare a 10-week program of resistance exercise plus creatine (EXSUPP) with resistance exercise alone (EXPLA), each with 20 participants.

DETAILED DESCRIPTION:
Colorectal cancer is the third most commonly diagnosed cancer in the world. Sarcopenia, defined as a loss of skeletal muscle mass and function, is highly prevalent in colorectal cancer, with rates of up to 60% reported. Sarcopenia etiology in cancer is multifactorial, with aging and inactivity compounded by treatment toxicities, malnutrition, tumor burden, and high-grade inflammation. Consequently, it's unlikely that unimodal interventions will be sufficient to overcome the burden of sarcopenia in this population. Creatine monohydrate is a naturally occurring compound in the body that plays a critical role in energy provision during exercise.4 Creatine is the most widely studied nutritional supplement to date, with well over 1,000 studies establishing its safety and effectiveness in men, women and older adults, in addition to other clinical populations. There is strong and consistent evidence that creatine supplementation can enhance the positive adaptations to resistance training in older adults and clinical populations. Therefore, there is strong potential for the application of creatine and resistance training to offset the decline in muscle mass and function after cancer treatment. The purpose of the proposed study is to examine the feasibility and acceptability of creatine supplementation combined with resistance exercise, compared to resistance exercise alone in individuals treated for colorectal cancer who are sarcopenic. We propose a randomized controlled pilot trial, examining the effects of 10-week multimodal resistance exercise and creatine supplementation (EXSUPP) (n=20) relative to resistance exercise alone (EXPLA) (n=20) in individuals treated for colorectal cancer who have sarcopenia. The specific aims of this project are to 1) determine the feasibility and acceptability of the intervention in colorectal cancer patients? diagnosed with sarcopenia after cancer treatment, 2) compare the effects of an exercise and creatine supplementation intervention (EXSUPP) to exercise alone (EXPLA) on body composition, muscle strength, physical function, and quality of life and 3) explore muscle molecular-level adaptations, i.e., mitochondrial health and protein turnover, in response to the interventions. This project will be one of the first to combine exercise with creatine, specifically targeting sarcopenia in individuals previously treated for colorectal cancer. This project is directly in line with the priority research initiative from the NCI Cancer MoonshotSM to "minimize Cancer Treatment's Debilitating Side Effects." Our trial is innovative in addressing one of the most important health problems for individuals treated for colorectal cancer in that it will be the first to 1) examine the feasibility and acceptability of a multimodal exercise and nutritional intervention relative to exercise alone in individuals treated for colorectal cancer who are sarcopenic and 2) explore the molecular mechanisms underpinning the response to exercise and nutritional interventions.

ELIGIBILITY:
Inclusion Criteria:

* . Individuals ≥12 months post treatment for colorectal cancer
* >18 years

Exclusion Criteria:

1. are receiving active treatment for their cancer;
2. have a any contraindication to exercise participation;
3. have been participating in structured resistance exercise 2 or more times per week for the past 6 months;
4. are currently taking supplements containing creatine for 4 weeks prior to the start of the RCT, or
5. are receiving medications that might alter body composition (metformin, corticosteroids etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 10-weeks
  Number of individuals enrolled across study timeframe
Retention | 10-weeks
  Proportion of individuals who return for follow-up testing
Supplementation Adherence | 10-weeks
  Proportion of daily supplementation taken
Exercise Adherence | 10-weeks
  Proportion of total exercise achieved

SECONDARY OUTCOMES:
Muscular Strength | 0 and 10-weeks
  Leg Press and Chest press 5 repetition maximum
Handgrip Strength | 0 and 10-weeks
  Handgrip Dynamometry (Jamar Plus+)
Body Composition | 0 and 10-weeeks
  DEXA
Physical Function | 0 and 10-weeks
  Short Physical Performance Battery
Health-Related Quality of Life | 0 and 10-weeks
  European Organization for Research and Treatment of Cancer QoL Questionnaire Core 30 (EORTC-QLQ-C30).
Sarcopenia related quality of life | 0 and 10-weeks
  Sarcopenia-related HRQOL will be assessed using a sarcopenia-specific questionnaire (SarQoL).
Inflammatory Markers | 0 and 10-weeks
  C reative protein, Interleukin 6 and Tumor necrosis factor alpha
Intramuscular Signaling and Mitochondrial Health and skeletal muscle regulation | 0 and 10-weeks
  Intramuscular markers of mitochondrial content and biogenesis (complex I-V content, citrate synthase activity, and PGC-1a protein expression)

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran Fairman, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States